CLINICAL TRIAL: NCT01301690
Title: Development of a Novel Methodology Using BMVC Staining as an Assistance to Cancer Cytological Diagnosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Li-Jen Liao, Department of Otolaryngology, Far Eastern Memorial Hospital
Other Study IDs: FEMH No.:98041-3
Record Dates: First submitted 2011-02-21; First posted 2011-02-23 (Estimated); Last update posted 2011-09-19 (Estimated); Status verified 2011-09

CONDITIONS: Neck Mass
Keywords: neck mass; ultrasound; FNA; BMVC

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Neck masses: Neck mass received US and US-FNA

SUMMARY:
3,6-bis(1-methyl-4-vinylpyridinium) carbazole diiodide (BMVC) is an inorganic chemical compound (Figure1). The uptake of BMVC in cancer cells and normal cells are different. Recently, a simple handheld device (Figure1) based on the fluorescence analysis of stained cells was established to instantly differentiate cancer cells from normal cells. The investigators want to quantitatively measure the fluorescence expression of BMVC in normal and cancer cells and explore the usefulness of this staining in head and neck lumps.

ELIGIBILITY:
Inclusion Criteria:

* patients (age range from 18 to 90 years old) with neck lumps, receiving sonographic examination and FNA cytologic study.

Exclusion Criteria:

* No cytology data

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We propose to collect consecutive patients (age range from 18 to 90 years old) with neck lumps, receiving sonographic examination and FNA cytologic study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-01

CONTACTS AND LOCATIONS:
Overall Officials: Li-Jen Liao, MD, Study Director — Department of Otolaryngology Far Eastern Memorial Hospital, Taipei, Taiwan
Locations (1):
- Department of Otolaryngology Far Eastern Memorial Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Liao LJ, Kang CC, Jan IS, Chen HC, Wang CL, Lou PJ, Chang TC. Improved diagnostic accuracy of malignant neck lumps by a simple BMVC staining assay. Analyst. 2009 Apr;134(4):708-11. doi: 10.1039/b814417f. Epub 2009 Jan 24. PMID 19305919